CLINICAL TRIAL: NCT01847560
Title: A Description of Warfarin and NOAC Utilization Patterns Including Initiation, Switching, and Discontinuation
Brief Title: Anticoagulant Utilization Pattern
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1160.177
Record Dates: First submitted 2013-04-18; First posted 2013-05-07 (Estimated); Results first posted 2019-06-27 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Dabigatran
- Warfarin or other New Oral Anticoagulant (NOAC)

SUMMARY:
This study plans to describe utilization patterns for oral anticoagulants over time in patients with non-valvular atrial fibrillation at risk for stroke using electronic claims data from a United States commercial insurance database.

ELIGIBILITY:
Inclusion criteria:

* A recorded diagnosis of atrial fibrillation
* Initiation of oral anticoagulant medication
* Congestive Heart Failure, Hypertension, Age > 75, Diabetes Mellitus, Prior Stroke or Transient Ischemic Attack, Vascular Disease, Age 65-74, Sex Category (CHA2DS2-VASc) Score >=1
* At least 18 years of age on the date of anticoagulant initiation

Exclusion criteria:

* Patients with missing or ambiguous age or sex information
* Patients with documented evidence of valvular disease
* Patients with less than 12 months enrolment in the UnitedHealth Research Database preceding the first dispensing
* Patients with prior use of any oral anticoagulant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age and older with non-valvular AF at risk for stroke treated with oral anticoagulation
Sampling Method: Non-Probability Sample
Enrollment: 333664 (Actual)
Dates: Start 2013-04-17 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study used a cohort design with descriptive analyses, using data from January 2009 through September 2015. The study was conducted within two US-based longitudinal healthcare claims databases (MarketScan and UnitedHealth Research Database).
Pre-assignment Details: The data source for this project was a combination of claims data from UnitedHealth, a commercial health insurer, and MarketScan, a research claims database from commercial employer-sponsored health plans both of which provide comprehensive medical coverage for members with active policies.
Groups:
- Cohort UnitedHealth Dabigatran Users: Patients with a diagnosis of non-valvular atrial fibrillation (NVAF) new initiators of Dabigatran who were enrolled for a minimum of 12 months in UnitedHealth cohort before treatment initiation.
- Cohort UnitedHealth Rivaroxaban Users: Patients with a diagnosis of non-valvular atrial fibrillation (NVAF) new initiators of Rivaroxaban who were enrolled for a minimum of 12 months in UnitedHealth cohort before treatment initiation.
- Cohort UnitedHealth Apixaban Users: Patients with a diagnosis of non-valvular atrial fibrillation (NVAF) new initiators of Apixaban who were enrolled for a minimum of 12 months in UnitedHealth cohort before treatment initiation.
- Cohort UnitedHealth WarfarinUsers (After Dabigatran Available): Patients with a diagnosis of non-valvular atrial fibrillation (NVAF) new initiators of Warfarin after Dabigatran became available who were enrolled for a minimum of 12 months in UnitedHealth cohort before treatment initiation.
- Cohort UnitedHealth WarfarinUsers(Before Dabigatran Available): Patients with a diagnosis of non-valvular atrial fibrillation (NVAF) new initiators of Warfarin before Dabigatran became available who were enrolled for a minimum of 12 months in UnitedHealth cohort before treatment initiation.
- Cohort MarketScan Dabigatran Users: Patients with a diagnosis of non-valvular atrial fibrillation (NVAF) new initiators of Dabigatran who were enrolled for a minimum of 12 months in MarketScan cohort before treatment initiation.
- Cohort MarketScan Rivaroxaban Users: Patients with a diagnosis of non-valvular atrial fibrillation (NVAF) new initiators of Rivaroxaban who were enrolled for a minimum of 12 months in MarketScan cohort before treatment initiation.
- Cohort MarketScan Apixaban Users: Patients with a diagnosis of non-valvular atrial fibrillation (NVAF) new initiators of Apixaban who were enrolled for a minimum of 12 months in MarketScan cohort before treatment initiation.
- Cohort MarketScan WarfarinUsers (After Dabigatran Available): Patients with a diagnosis of non-valvular atrial fibrillation (NVAF) new initiators of Warfarin after Dabigatran became available who were enrolled for a minimum of 12 months in MarketScan cohort before treatment initiation.
- Cohort MarketScan WarfarinUsers(Before Dabigatran Available): Patients with a diagnosis of non-valvular atrial fibrillation (NVAF) new initiators of Warfarin before Dabigatran became available who were enrolled for a minimum of 12 months in MarketScan cohort before treatment initiation.
Period: Overall Study
Arm/Group | Cohort UnitedHealth Dabigatran Users | Cohort UnitedHealth Rivaroxaban Users | Cohort UnitedHealth Apixaban Users | Cohort UnitedHealth WarfarinUsers (After Dabigatran Available) | Cohort UnitedHealth WarfarinUsers(Before Dabigatran Available) | Cohort MarketScan Dabigatran Users | Cohort MarketScan Rivaroxaban Users | Cohort MarketScan Apixaban Users | Cohort MarketScan WarfarinUsers (After Dabigatran Available) | Cohort MarketScan WarfarinUsers(Before Dabigatran Available)
Started | 13464 | 19955 | 9731 | 56655 | 27731 | 28343 | 40971 | 19829 | 77547 | 39438
Completed | 13464 | 19955 | 9731 | 56655 | 27731 | 28343 | 40971 | 19829 | 77547 | 39438
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients with nonvalvular atrial fibrillation at risk for stroke initiating oral anticoagulants and a description of existing utilization patterns for warfarin and for the new oral anticoagulant (NOAC) medications as they become available over time.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort UnitedHealth Dabigatran Users | Cohort UnitedHealth Rivaroxaban Users | Cohort UnitedHealth Apixaban Users | Cohort UnitedHealth WarfarinUsers (After Dabigatran Available) | Cohort UnitedHealth WarfarinUsers(Before Dabigatran Available) | Cohort MarketScan Dabigatran Users | Cohort MarketScan Rivaroxaban Users | Cohort MarketScan Apixaban Users | Cohort MarketScan WarfarinUsers (After Dabigatran Available) | Cohort MarketScan WarfarinUsers(Before Dabigatran Available) | Total
Number analyzed (Participants) | 13464 | 19955 | 9731 | 56655 | 27731 | 28343 | 40971 | 19829 | 77547 | 39438 | 333664
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.07 (11.4) | 70.04 (11.45) | 72.18 (11.05) | 73.64 (10.28) | 71.7 (10.8) | 67.17 (12.11) | 67.63 (12.21) | 69.42 (12.32) | 71.03 (12.11) | 69.1 (12.4) | 70.4 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5017 | 7939 | 4225 | 24620 | 11699 | 10096 | 15305 | 7776 | 30293 | 15539 | 132509
  Male | 8447 | 12016 | 5506 | 32035 | 16032 | 18247 | 25666 | 12053 | 47254 | 23899 | 201155
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Description of the Characteristics of Anticoagulant Initiators
Description: The analyses described the characteristics of patients treated with various oral anticoagulants. CHA2DS2-VASc stroke risk score is calculated based on the following conditions: Congestive heart failure/ Left ventricular (LV) dysfunction, Hypertension, Age (≥ 75), Diabetes Mellitus, Stroke/ transient ischemic attack (TIA) /thromboembolism, Vascular disease, Age 65-74, female gender. HAS-BLED bleeding risk score is calculated based on the following conditions: Hypertension, Abnormal renal and liver function, Stroke (1 point), Bleeding history or predisposition, Labile international normalized ratio (INR), Elderly (>65 years), Drugs and Alcohol. CHA2DS2-VASc stroke risk score may range from 0 to 9 with 0 being the best outcome. HAS-BLED bleeding risk score may range from 0 to 9 with 0 being the best outcome. New initiators of warfarin before Dabigatran became available were only characterized in terms of age and sex (results provided above).
Time Frame: From January 2009 to September 2015 (The study period)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Cohort UnitedHealth Warfarin Users: Patients with a diagnosis of non-valvular atrial fibrillation (NVAF) new initiators of Warfarin after Dabigatran became available who were enrolled for a minimum of 12 months in UnitedHealth cohort before treatment initiation.
- Cohort MarketScan Warfarin Users: Patients with a diagnosis of non-valvular atrial fibrillation (NVAF) new initiators of Warfarin after Dabigatran became available who were enrolled for a minimum of 12 months in MarketScan cohort before treatment initiation.
Arm/Group | Cohort UnitedHealth Dabigatran Users | Cohort UnitedHealth Warfarin Users | Cohort UnitedHealth Rivaroxaban Users | Cohort UnitedHealth Apixaban Users | Cohort MarketScan Dabigatran Users | Cohort MarketScan Warfarin Users | Cohort MarketScan Rivaroxaban Users | Cohort MarketScan Apixaban Users
Number analyzed (Participants) | 13464 | 56655 | 19955 | 9731 | 28343 | 77547 | 40971 | 19829
Scores on a scale
  CHA2DS2-VASc score | 3.41 (1.73) | 4.30 (1.75) | 3.59 (1.75) | 3.82 (1.72) | 2.92 (1.58) | 3.62 (1.69) | 3.12 (1.68) | 3.34 (1.73)
  HAS-BLED score | 2.52 (1.15) | 2.91 (1.18) | 2.63 (1.15) | 2.76 (1.16) | 2.18 (1.02) | 2.51 (1.12) | 2.32 (1.1) | 2.47 (1.14)

2. Primary Outcome: Percentage of Patients Initiating Specific Anticoagulant
Description: Proportion of patients initiating specific anticoagulant over time per arm in source cohort is estimated and is expressed in percentage. This is related to UnitedHealth database and no treatment initiation rate was estimated in MarketScan as the study cohort was defined from a population of oral anticoagulants users. The overall number of participants analyzed "609201" reported for each of the treatment arm below corresponds to overall patients numbers in UnitedHealth for the entire study period rather than for each of the treatment arm. Likewise the number of participants for each of the treatment arm for different time period corresponds to the total number of participants for the specific study period rather than for each of the treatment arm. Incident users at given time period could also be counted in later time period if the patient discontinued the drug and had re-entry during the study period.
Time Frame: From January 2009 to September 2015 (The study period)
Population: Source cohort in a calendar time window includes all patients with at least one day eligibility. A random date within the time window selected and set as the index date. Patients dispensed of an anticoagulant before assigned index date will be removed, unless they are identified as new initiators for that particular time period.
Measure: Number; unit: Percentage of initiators (%)
Groups:
- Warfarin Users: Patients with a diagnosis of non-valvular atrial fibrillation (NVAF) initiating treatment with Warfarin in source cohort.
- Dabigatran Users: Patients with a diagnosis of non-valvular atrial fibrillation (NVAF) initiating treatment with Dabigatran in source cohort.
- Rivaroxaban Users: Patients with a diagnosis of non-valvular atrial fibrillation (NVAF) initiating treatment with Rivaroxaban in source cohort.
- Apixaban Users: Patients with a diagnosis of non-valvular atrial fibrillation (NVAF) initiating treatment with Apixaban in source cohort.
Arm/Group | Warfarin Users | Dabigatran Users | Rivaroxaban Users | Apixaban Users
Number analyzed (Participants) | 609201 | 609201 | 609201 | 609201
Percentage of initiators (%)
  January 2009 - September2010: number analyzed (Participants) | 72574 | 72574 | 72574 | 72574
  January 2009 - September2010 | 15.7 | NA — No treatment initiation during this period | NA — No treatment initiation during this period | NA — No treatment initiation during this period
  October2010 - June2011: number analyzed (Participants) | 67422 | 67422 | 67422 | 67422
  October2010 - June2011 | 5.4 | 2.1 | NA — No treatment initiation during this period | NA — No treatment initiation during this period
  July2011 -Dec 2011: number analyzed (Participants) | 66458 | 66458 | 66458 | 66458
  July2011 -Dec 2011 | 2.9 | 2.2 | NA — No treatment initiation during this period | NA — No treatment initiation during this period
  January2012-June2012: number analyzed (Participants) | 64745 | 64745 | 64745 | 64745
  January2012-June2012 | 3.4 | 1.9 | 1.5 | NA — No treatment initiation during this period
  July2012-December2012: number analyzed (Participants) | 55742 | 55742 | 55742 | 55742
  July2012-December2012 | 2.9 | 1.3 | 1.5 | NA — No treatment initiation during this period
  January2013-June2013: number analyzed (Participants) | 51641 | 51641 | 51641 | 51641
  January2013-June2013 | 2.3 | 0.8 | 1.8 | 0.3
  July2013-December2013: number analyzed (Participants) | 52563 | 52563 | 52563 | 52563
  July2013-December2013 | 2.0 | 0.6 | 1.9 | 0.7
  January2014-June2014: number analyzed (Participants) | 46437 | 46437 | 46437 | 46437
  January2014-June2014 | 1.7 | 0.5 | 2.2 | 1.0
  July2014-December2014: number analyzed (Participants) | 45483 | 45483 | 45483 | 45483
  July2014-December2014 | 1.6 | 0.4 | 2.0 | 1.3
  January2015-June2015: number analyzed (Participants) | 43806 | 43806 | 43806 | 43806
  January2015-June2015 | 1.6 | 0.3 | 2.0 | 1.7
  July2015-September2015: number analyzed (Participants) | 42330 | 42330 | 42330 | 42330
  July2015-September2015 | 0.7 | 0.1 | 1.0 | 1.0

3. Primary Outcome: Percentage of Patients Initiating Specific Anticoagulant Dose - Dabigatran
Description: Percentage of patients initiating specific anticoagulant dose of dabigatran across all time periods combined in the unmatched cohort for UnitedHealth and MarketScan cohort are presented. Proportion of patients initiating specific anticoagulant over time per arm in source cohort is estimated and is expressed in percentage.
Time Frame: From January 2009 to September 2015 (The study period)
Population: Patients initiating treatment in source cohort.
Measure: Number; unit: Percentage of initiators (%)
Groups:
- Cohort UnitedHealth Dabigatran Users: Patients with a diagnosis of non-valvular atrial fibrillation (NVAF) initiating treatment with dabigatran in UnitedHealth cohort.
- Cohort MarketScan Dabigatran Users: Patients with a diagnosis of non-valvular atrial fibrillation (NVAF) initiating treatment with dabigatran in MarketScan cohort.
Arm/Group | Cohort UnitedHealth Dabigatran Users | Cohort MarketScan Dabigatran Users
Number analyzed (Participants) | 13464 | 28343
Percentage of initiators (%)
  150 milligram (mg) | 90.7 | 90.7
  75 mg | 9.3 | 9.3

4. Primary Outcome: Percentage of Patients Initiating Specific Anticoagulant Dose - Apixaban
Description: Percentage of patients initiating specific anticoagulant dose of apixaban across all time periods combined in the unmatched cohort for UnitedHealth and MarketScan cohort are presented. Proportion of patients initiating specific anticoagulant over time per arm in source cohort is estimated and is expressed in percentage.
Time Frame: From January 2009 to September 2015 (The study period)
Population: Patients initiating treatment in source cohort.
Measure: Number; unit: Percentage of initiators (%)
Groups:
- Cohort UnitedHealth Apixaban Users: Patients with a diagnosis of non-valvular atrial fibrillation (NVAF) initiating treatment with apixaban in UnitedHealth cohort.
- Cohort MarketScan Apixaban Users: Patients with a diagnosis of non-valvular atrial fibrillation (NVAF) initiating treatment with apixaban in MarketScan cohort.
Arm/Group | Cohort UnitedHealth Apixaban Users | Cohort MarketScan Apixaban Users
Number analyzed (Participants) | 9731 | 19829
Percentage of initiators (%)
  5 mg | 82.4 | 84.4
  2.5 mg | 17.6 | 15.6

5. Primary Outcome: Percentage of Patients Initiating Specific Anticoagulant Dose - Rivaroxaban
Description: Percentage of patients initiating specific anticoagulant dose of rivaroxaban across all time periods combined in the unmatched cohort for UnitedHealth and MarketScan cohort are presented. Proportion of patients initiating specific anticoagulant over time per arm in source cohort is estimated and is expressed in percentage.
Time Frame: From January 2009 to September 2015 (The study period)
Population: Patients initiating treatment in source cohort.
Measure: Number; unit: Percentage of initiators (%)
Groups:
- Cohort UnitedHealth Rivaroxaban Users: Patients with a diagnosis of non-valvular atrial fibrillation (NVAF) initiating treatment with rivaroxaban in UnitedHealth cohort.
- Cohort MarketScan Rivaroxaban Users: Patients with a diagnosis of non-valvular atrial fibrillation (NVAF) initiating treatment with rivaroxaban in MarketScan cohort.
Arm/Group | Cohort UnitedHealth Rivaroxaban Users | Cohort MarketScan Rivaroxaban Users
Number analyzed (Participants) | 19955 | 40971
Percentage of initiators (%)
  20 mg | 74.0 | 76.4
  15 mg | 18.4 | 16.7
  10 mg | 7.6 | 7.0

6. Secondary Outcome: Treatment Persistence Over Time
Description: Overall treatment persistence in UnitedHealth and MarketScan cohorts are presented as the percentage of patients who were persistent to treatment after 3, 6 and 12 months of follow-up for all time periods combined and matched cohort. Based on two US-based longitudinal healthcare claims databases (MarketScan and unitedHealth Research Database) the three separate study cohorts warfarin vs dabigatran, warfarin vs rivaroxaban and warfarin vs apixaban cohort were formed for each database.
Time Frame: From January 2009 to September 2015 (The study period)
Population: Patients were matched within calendar quarters (3 months period) the various NOACs were individually matched to warfarin on an exposure propensity score (PS) in a 1:1 fixed ratio using a nearest neighbor technique and a caliper of 0.05.
Measure: Number; unit: Percentage of participants (%)
Groups:
- Cohort UnitedHealth Dabigatran (Dabigatran vs Warfarin); Cohort MarketScan Dabigatran (Dabigatran vs Warfarin): Patients exposed to dabigatran were matched to warfarin on an exposure propensity score (PS) on a 1:1 fixed ratio using a nearest neighbor technique and a caliper of 0.05.
- Cohort UnitedHealth Warfarin (Warfarin vs Dabigatran); Cohort MarketScan Warfarin (Warfarin vs Dabigatran): Patients exposed to warfarin were matched to dabigatran on an exposure propensity score (PS) on a 1:1 fixed ratio using a nearest neighbor technique and a caliper of 0.05.
- Cohort Unitedhealth Rivaroxaban (Rivaroxaban vs Warfarin); Cohort MarketScan Rivaroxaban (Rivaroxabna vs Warfarin): Patients exposed to rivaroxaban were matched to warfarin on an exposure propensity score (PS) on a 1:1 fixed ratio using a nearest neighbor technique and a caliper of 0.05.
- Cohort Unitedhealth Warfarin (Warfarin vs Rivaroxaban); Cohort MarketScan Warfarin (Warfarin vs Rivaroxaban): Patients exposed to warfarin were matched to rivaroxaban on an exposure propensity score (PS) on a 1:1 fixed ratio using a nearest neighbor technique and a caliper of 0.05.
- Cohort Unitedhealth Apixaban (Apixaban vs Warfarin); Cohort MarketScan Apixaban (Apixaban vs Warfarin): Patients exposed to apixaban were matched to warfarin on an exposure propensity score (PS) on a 1:1 fixed ratio using a nearest neighbor technique and a caliper of 0.05.
- Cohort Unitedhealth Warfarin (Warfarin vs Apixaban); Cohort MarketScan Warfarin (Warfarin vs Apixaban): Patients exposed to warfarin were matched to apixaban on an exposure propensity score (PS) on a 1:1 fixed ratio using a nearest neighbor technique and a caliper of 0.05.
Arm/Group | Cohort UnitedHealth Dabigatran (Dabigatran vs Warfarin) | Cohort UnitedHealth Warfarin (Warfarin vs Dabigatran) | Cohort Unitedhealth Rivaroxaban (Rivaroxaban vs Warfarin) | Cohort Unitedhealth Warfarin (Warfarin vs Rivaroxaban) | Cohort Unitedhealth Apixaban (Apixaban vs Warfarin) | Cohort Unitedhealth Warfarin (Warfarin vs Apixaban) | Cohort MarketScan Dabigatran (Dabigatran vs Warfarin) | Cohort MarketScan Warfarin (Warfarin vs Dabigatran) | Cohort MarketScan Rivaroxaban (Rivaroxabna vs Warfarin) | Cohort MarketScan Warfarin (Warfarin vs Rivaroxaban) | Cohort MarketScan Apixaban (Apixaban vs Warfarin) | Cohort MarketScan Warfarin (Warfarin vs Apixaban)
Number analyzed (Participants) | 11927 | 11927 | 15522 | 15522 | 7712 | 7712 | 24141 | 24141 | 26066 | 26066 | 12578 | 12578
Percentage of participants (%)
  After 3 months of follow-up | 52.19 | 52.86 | 53.17 | 51.58 | 51.84 | 48.29 | 57.92 | 53.25 | 58.33 | 53.27 | 58.24 | 51.17
  After 6 months of follow-up | 30.96 | 28.16 | 31.53 | 26.11 | 27.71 | 21.68 | 33.09 | 26.78 | 35.49 | 25.83 | 33.25 | 23.11
  After 12 months of follow-up | 15.07 | 11.86 | 13.54 | 9.63 | 9.14 | 5.56 | 15.47 | 10.18 | 16.50 | 8.93 | 13.20 | 6.22

ADVERSE EVENTS:
Time Frame: Safety related information was not captured during this study.
Description: This was an observational study based on existing data (secondary data use); all patient data are de-identified and analyzed in aggregate. Individual patient safety related information was not designed to assess for this study; therefore the individual safety reporting was not applicable for this study.
Arm/Group | Cohort UnitedHealth Dabigatran Users | Cohort UnitedHealth Rivaroxaban Users | Cohort UnitedHealth Apixaban Users | Cohort UnitedHealth WarfarinUsers (After Dabigatran Available) | Cohort UnitedHealth WarfarinUsers(Before Dabigatran Available) | Cohort MarketScan Dabigatran Users | Cohort MarketScan Rivaroxaban Users | Cohort MarketScan Apixaban Users | Cohort MarketScan WarfarinUsers (After Dabigatran Available) | Cohort MarketScan WarfarinUsers(Before Dabigatran Available)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-07-31): https://cdn.clinicaltrials.gov/large-docs/60/NCT01847560/Prot_SAP_000.pdf